CLINICAL TRIAL: NCT02960633
Title: Direct Anterior Approach (DAA) for Total Hip Arthroplasty (THA): Corail Prosthesis With or Without Collar Design
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ZOL (Other)
Responsible Party: Principal Investigator, Jens Vanbiervliet, Resident orthopedic Surgery, ZOL
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/073U
Record Dates: First submitted 2016-11-03; First posted 2016-11-09 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Coxarthritis

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- THA with Collar (Active Comparator): THA with Collar
  Interventions: Device: Corail with collar.
- THA without Collar (Active Comparator): THA without Collar
  Interventions: Device: Corail without collar.

INTERVENTIONS:
Device: Corail with collar.
  Arms: THA with Collar
Device: Corail without collar.
  Arms: THA without Collar

SUMMARY:
Direct Anterior Approach (DAA) for Total Hip Arthroplasty (THA): Corail prosthesis with or without collar design. Randomized study design focusing on radiolucent lines on standard x-ray.

ELIGIBILITY:
Inclusion Criteria:

* primary THA

Exclusion Criteria:

* fractured hips

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
The investigators will measure radiolucent lines on X-ray. | 5 year
  Hypothesis: Collar shows more radiolucent lines on xray in Gruen zone 7.